CLINICAL TRIAL: NCT06623825
Title: Evaluating the Efficiency of Smart Glasses in Reducing Patient Care Time in Emergency Medicine: Evidence From the Hangzhou Asian Games
Brief Title: Smart Glasses in Emergency Medicine From the Hangzhou Asian Games
Acronym: SGINHZAG
Status: Completed | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yucai Hong, Head of Emergency Department, Sir Run Run Shaw Hospital
Other Study IDs: v1.020230801
Record Dates: First submitted 2024-09-14; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Trauma Injury; Acute Coronary Syndrome; Stroke, Acute; Septic Shock
Keywords: Telemedicine; Tele-consultation; Smart glasses; Emergency Medicine
MeSH Terms: conditions — Accidental Injuries; Acute Coronary Syndrome; Stroke; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARTS: the teleconsultation by AR telemedicine system group
  Interventions: Device: teleconsultation by Augmented Reality smart glasses
- non-ARTS: no teleconsultation by AR telemedicine system groups,but by the traditional methods like radios, telephonecalls
  Interventions: Device: teleconsultation by two-way radio connection.

INTERVENTIONS:
Device: teleconsultation by Augmented Reality smart glasses — The device operated on Android 9.0 and it connected to 5G connection with a bandwidth speed 30-mbps delivering a very low latency. The device supported real time screen sharing and therefore the data were collected from smart glasses including visual and audio with real-time two-way communications. Physicians at the hospital can access the information and video via a mobile app, enabling continuous monitoring of patients. The features facilitate healthcare providers at SRRSH and medical personnel in the HAG2022 polyclinic to discuss the patient's condition, exchange, and deliberate on the pre-hospital medical examinations of the patient.
  Other Names: realtime teleconsultation by Augmented Reality smart glasses
  Groups: ARTS
Device: teleconsultation by two-way radio connection. — adhering to the standard conventional triage process without the AR tool, only using a two-way radio connection.
  Other Names: the traditional teleconsultation by two-way radio connection.
  Groups: non-ARTS

SUMMARY:
The findings of our study will reveal that using smart glasses in the emergency department(ED) could facilitate patient admission. AR Smart Glasses offer the potential to enhance the effectiveness and speed of treatment within ED.

DETAILED DESCRIPTION:
Study Design:

This study will be conducted at Sir Run Run Shaw Hospital (SRRSH), China. This study aims to compare the outcomes of two groups: the intervention group, utilizing the Augmented Reality (AR) smart glasses, and the control group, adhering to the standard conventional triage process without the AR tool, only using a two-way radio connection.

Augmented Reality tool The AR tool used in this study will be a smart glasses manufactured by Rokid AR Studio(Hangzhou, China). It was Rokid glass 2 model released in 2020. The device operated on Android 9.0 and it connected to 5G connection with a bandwidth speed 30-mbps delivering a very low latency. The device supported real time screen sharing and therefore the data were collected from smart glasses including visual and audio with real-time two-way communications. Physicians at the hospital can access the information and video via a mobile app, enabling continuous monitoring of patients. The features facilitate healthcare providers at SRRSH and medical personnel in the HAG2022 polyclinic to discuss the patient's condition, exchange, and deliberate on the pre-hospital medical examinations of the patient.

Participants:

The study, will be conducted between September 13, 2023, and October 28, 2023, included the recruitment of all patients (older than 16 years old) presenting with acute illnesses who were admitted to the ED of SRRSH from the HAG2022 village polyclinic or the field of injury.

The Cases with incomplete data and cases where the patients would be not found will be excluded from this study. Cases involving technical difficulties encountered by operators using augmented reality (AR) smart glasses and loss of internet connection will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with acute illnesses like acute coronary syndrome，acute sepsis，stroke，trauma who will be admitted to the ED of SRRSH from the HAG2022 village polyclinic or the field of injury.

Exclusion Criteria:

* The Cases with incomplete data and cases where the patients will be not found will be excluded from this study. Cases involving technical difficulties encountered by operators using augmented reality (AR) smart glasses and loss of internet connection will be excluded from the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Following the completion of the research period, there will be 80 patients categorized into the ARTS cohort consisting of 10 patients and the non-ARTS cohort comprising 70 patients. Gender and age demographics for ARTS and non-ARTS cohorts will be shown with no significant gender differences.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
the consult response time (CRT) | through study completion, an average of 1 year
  CRT refers to the duration from when consulting physicians are called to evaluate patients in the ED to their response
pre-preparation time (PPT ) | through study completion, an average of 1 year
  PPT refers to the duration required to prepare the patient for subsequent management

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No